CLINICAL TRIAL: NCT04224376
Title: Improving Maximal Strength in the Initial Postoperative Phase After Anterior Cruciate Ligament Reconstruction Surgery: Randomized Controlled Trial of an App-Based Serious Gaming Approac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Clausen, Jan-Dierk Dr., Principal Investigator, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3102-2016 VKB
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: ACL rupture; return to sports
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation (No Intervention): Normal postoperative treatment protocol with physiotherapy after ACL surgery
- Serious Gaming (Experimental): In the training group each patient was additionally provided with a GenuSport knee trainer device (prototype plus tablet with software application) with the active knee extension training program for 6 weeks. Other postoperative treatment was identical.
  Interventions: Device: App based Serious Gaming with the Genu Sport knee trainer

INTERVENTIONS:
Device: App based Serious Gaming with the Genu Sport knee trainer — The Genu Sport knee trainer has a strength monitoring unit with three integrated sensors which is placed in the popliteal area and a tablet with the application which allows to transfer the raised force into the game modus. Each training session in our study takes around 5 minutes and is performed autonomously by the patient in his bed with 45° degrees of upper body evaluation while the patient holds the tablet in both hands. By simply pushing his knee downward onto the measuring unit the patient can apply the force.
  Arms: Serious Gaming

SUMMARY:
The investigators designed a prospective randomized trial to evaluate whether an app based active muscle training program (GenuSport) can improve the postoperative strength by starting rehabilitation immediately after primary anterior cruciate ligament (ACL) reconstruction surgery as already shown for patients who underwent total knee arthroplasty. To the investigators knowledge this is the first study analyzing immediate postoperative serious gaming based training with the GenuSport device based on strength improvement.

DETAILED DESCRIPTION:
The study is designed as a prospective randomized control trial. Participants awaiting primary ACL reconstruction surgery were recruited at a single tertiary healthcare center between April 2016 and February 2018. An ethical approval has been given by MHH ethic committee and an IRB was involved. Due to different postoperative treatment protocols and different surgical approaches we could include participants between 13 and 46 years. A computer based randomization was performed by generating a list of randomized numbers which have been provided in sealed envelopes by an independent examiner. The postoperative treatment protocol was apart from the use of the GenuSport knee trainer identically standardized. The pain management was the same for all patients, none of the participants received a continuous peripheral nerve block. The postoperative physiotherapy protocol included gait training, assisted walking with crutches, active and passive knee mobilization, strength exercises and stair climbing. In the training group each participant was additionally provided with a GenuSport knee trainer device (prototype plus tablet with software application) with the active knee extension training program for 6 weeks. Except of that fact the postoperative protocol was identical in both groups. Participant had to train five times daily with the knee trainer starting at the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients awaiting primary ACL reconstruction surgery
* Willingness to participate
* Ability to work with an app based training device

Exclusion Criteria:

* Additional meniscal suturing
* Additional collateral ligament repair
* Additional regenerative cartilage treatment
* Unwillingness to participate in the study

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Absolute and relative change in maximum strength | 6 weeks
  Primarily, change in maximum strength was analyzed both, as an absolute difference between week 6 and pre-surgery value (6 weeks - pre-surgery) and as a relative change (6 weeks / pre-surgery).

SECONDARY OUTCOMES:
Change in clinical outcome | 6 weeks
  IKDC, Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms)
Change in clinical outcome | 6 weeks
  KOOS
Change in clinical outcome | 6 weeks
  Tegner activity scale, scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer
Change in clinical outcome | 6 weeks
  Lysholm, Maximum 100 points higher score means better Outcome
Change in clinical outcome | 6 weeks
  VAS score, Values 0 to 10 higher values mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sanjay Weber-Spickschen, MD, Principal Investigator — Trauma Departement, Hanover Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frobell RB, Roos EM, Roos HP, Ranstam J, Lohmander LS. A randomized trial of treatment for acute anterior cruciate ligament tears. N Engl J Med. 2010 Jul 22;363(4):331-42. doi: 10.1056/NEJMoa0907797. PMID 20660401
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Sims J, Cosby N, Saliba EN, Hertel J, Saliba SA. Exergaming and static postural control in individuals with a history of lower limb injury. J Athl Train. 2013 May-Jun;48(3):314-25. doi: 10.4085/1062-6050-48.2.04. Epub 2013 Feb 20. PMID 23675790
- [Background] Horstmann H, Krost E, Welke B, Kerling A, Hanke A, Jakubowitz E, Weber-Spickschen TS. The determination of the validity of an application-based knee-training device. Assist Technol. 2019;31(5):259-266. doi: 10.1080/10400435.2018.1441924. Epub 2018 Apr 10. PMID 29465298